CLINICAL TRIAL: NCT03661606
Title: Measuring the Effect of High Altitude (Hypoxia) on an Individual's Physiology - an Analytical Study to Validate the Performance of the Biovitals™ Analytics Engine (BA Engine - Altitude Study)
Brief Title: Biovitals Analytics Engine - Altitude Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biofourmis Singapore Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PIEC/2018/013
Record Dates: First submitted 2018-09-01; First posted 2018-09-07 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring arm (Experimental): Subjects will wear one armband linked biosensor: the Everion® CD, to capture their HR, RR and activity levels, continuously for 4 days.
  Interventions: Other: Simulated Altitude Chamber

INTERVENTIONS:
Other: Simulated Altitude Chamber — Subjects will wear one armband linked biosensor: the Everion® CD, to capture their HR, RR and activity levels, continuously for 4 days.
  Measurements will be taken at sea level (baseline), during controlled rest and normal day-to-day activities without exercise for the first 3 days to establish an individual's physiological baseline. On Day 4 subjects will be monitored for another period of controlled rest followed by 2 hours in a simulated altitude (intervention) chamber with altitude change of 3000 meters. At the chamber site, subject will rest quietly for 1 hour outside the chamber prior to entering the chamber for 2 hours. In the chamber, subjects will be asked to remain seated. At the completion of the chamber run, subjects will hand back the device and smartphone and complete a user experience survey. A follow up phone call to check on subjects will then be done on day 5 before closing the study.

SUMMARY:
Unexpected adverse health events resulting in a hospital admission can be potentially avoided by leveraging novel physiological sensors combined with advanced computational techniques to predict changes in physiology prior to the onset of symptoms. In other words, significant improvement in the prevention of avoidable hospitalization can be achieved via early detection and actionable insights of clinical deterioration at the individual patient level as they go about their normal day to day activities. Physiological changes can be a warning sign that a person's health is deteriorating and as such is an important component of an early detection tool.

The Biovitals Analytics Engine (BA Engine) is intended to be used with data from already validated sensors measuring physiological parameters, including heart rate (HR), respiratory rate (RR) and activity in ambulatory patients being monitored in a healthcare facility or at home. The device provides a continuous output- Biovitals™ Index (BI) which indicates whether the relationships among the patients monitored vital signs change from those measured at baseline (derived from measurements previously obtained during daily routine activities). The BI is based on an integrated computation evaluating changes in the parameters and their relationship to each other.

As part of the clinical validation of the BA Engine, it is important to first undertake an analytical validation to demonstrate that the BA correctly processes the physiological data for which it is designed, and generates an accurate detection of physiological change. In order to generate a measurable physiological change, subjects will move from sea level to an altitude environment which is known to cause increases in HR and RR.

DETAILED DESCRIPTION:
Subjects will wear one armband linked biosensor: the Everion® CD, to capture their HR, RR and activity levels, continuously for 4 days.

Measurements will be taken at sea level (baseline), during controlled rest and normal day-to-day activities without exercise for the first 3 days to establish an individual's physiological baseline. On Day 4 subjects will be monitored for another period of controlled rest followed by 2 hours in a simulated altitude (intervention) chamber with an altitude change of 3000 meters. At the chamber site, the subject will rest quietly for 1 hour outside the chamber prior to entering the chamber for 2 hours. In the chamber, subjects will be asked to remain seated. At the completion of the chamber run, subjects will hand back the device and smartphone and complete a user experience survey. A follow-up phone call to check on subjects will then be done on day 5 before closing the study.

ELIGIBILITY:
Inclusion Criteria:

* 50 Male or female, voluntary adults aged between ≥ 18 to ≤ 65 years
* Ability to read and understand basic English Language
* Women who are of childbearing potential, must if sexually active, agree to use appropriate contraceptive measures for the duration of the study
* Able to perform all activities in the study procedure

Exclusion Criteria:

* High altitude residents (>500m)
* Anemic
* Athlete
* Lung, airways and/or sinus pathology
* Previous myocardial infarction or coronary revascularization (PCI or CABG)
* Any prior history of heart failure
* Any prior history of moderate or severe valvular heart disease
* Any history of pulmonary disease (asthma, emphysema/ COPD, pulmonary hypertension)
* Any other medical condition or functional problems (e.g. previous intolerance or current contraindication to altitude, unable to exercise, skin problems, schizophrenia and bipolar disorder) that in the judgment of the investigator will impair the subjects ability to complete the processes needed in the clinical study
* Unable or unwillingness to sign the informed consent
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Analytical validation testing of the BA Engine's output | Changes in subjects physiology at an altitude of 3000m compared to baseline physiology
  This study aims to demonstrate that the BA Engine correctly processes monitored physiological data to generate accurate, reliable and precise detection of changes in an individual's physiology at high altitude (3000m) when compared to their baseline physiology at sea-level, as per its design specifications and to meet its intended use.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Aeromedical Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No